CLINICAL TRIAL: NCT07396337
Title: A Multicenter, Randomized, Double-Blind, Placebo-Controlled, Phase IIb Clinical Trial of QHRD106 Injection for the Treatment of Acute Ischemic Stroke
Brief Title: Study to Assess the Efficacy and Safety of QHRD106 Injection in Acute Ischemic Stroke.
Status: Recruiting | Phase: Phase 2 | Type: Interventional
Sponsor: Changzhou Qianhong Bio-pharma Co., Ltd. (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: PR-QHRD-106-ⅡB
Record Dates: First submitted 2026-02-01; First posted 2026-02-09 (Actual); Last update posted 2026-02-09 (Actual); Status verified 2026-02

CONDITIONS: Acute Ischemic Stroke
MeSH Terms: conditions — Ischemic Stroke | interventions — Population Groups

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (4):
- QHRD106 injection（Low-dose group） (Experimental)
  Interventions: Drug: QHRD106 Injection (Low-dose group)
- QHRD106 injection（Middle-dose group） (Experimental)
  Interventions: Drug: QHRD106 Injection (Middle-dose group)
- QHRD106 injection（High-dose group） (Experimental)
  Interventions: Drug: QHRD106 Injection (High-dose group)
- Placebo (Placebo Comparator)
  Interventions: Drug: Placebo

INTERVENTIONS:
Drug: QHRD106 Injection (Low-dose group) — Participants will receive QHRD106 injection (5600 IU) every 7 days with a total of 3 doses.
  Arms: QHRD106 injection（Low-dose group）
Drug: QHRD106 Injection (Middle-dose group) — Participants will receive QHRD106 injection (8400 IU) every 7 days with a total of 3 doses.
  Arms: QHRD106 injection（Middle-dose group）
Drug: QHRD106 Injection (High-dose group) — Participants will receive QHRD106 injection (12600 IU) every 7 days with a total of 3 doses.
  Arms: QHRD106 injection（High-dose group）
Drug: Placebo — Participants will receive placebo every 7 days with a total of 3 doses.
  Arms: Placebo

SUMMARY:
The purpose of this study is to determine the efficacy and safety of QHRD106 injection in treating acute ischemic stroke.

DETAILED DESCRIPTION:
This is a multicenter, randomized, double-blind, placebo-controlled, phase IIb clinical trial of QHRD106 injection for the treatment of acute ischemic stroke. The goal of this trial is to explore the efficacy and safety of different doses of QHRD106 injection in patients with acute ischemic stroke (AIS) who are unfit for reperfusion therapy within 24 hours of symptom onset.Participants will receive a low-dose QHRD106 injection (5600 IU), a middle-dose QHRD106 injection (8400 IU), a high-dose QHRD106 injection (12600 IU), or a placebo intravenously within 24 hours of stroke onset. They will be treated once every 7 days, with a total of 3 doses over the course of the study.

ELIGIBILITY:
Inclusion Criteria:

1. Age ≥ 18 years old and ≤ 80 years old;
2. Patients diagnosed as acute ischemic stroke according to the latest guidelines；
3. Patients who have not received or have no plan to receive standard intravenous thrombolysis within 24 hours after the onset of the disease and can complete the first administration of the investigational drug within 24 hours after the onset.；
4. Total National Institute of Health stroke scale (NIHSS)≥6 and ≤20, and the sum of NIHSS score for the upper limb and the lower limb is greater than or equal to 2；
5. The mRS score before the onset of the disease is ≤ 1 point;
6. Obtain the informed consent form signed by the patient or their guardian.

Exclusion Criteria:

1. Combine intracranial hemorrhagic diseases, including hemorrhagic stroke, epidural hematoma, intracranial hematoma, ventricular hemorrhage, subarachnoid hemorrhage, etc；
2. Individuals with any of the following allergy histories must be excluded: 1) Those who are allergic to the test drug or similar components; 2) Those who are allergic to the materials used in imaging examinations; 3) Those who are allergic to any drugs, medical devices, or products derived from pigs or other mammals (such as porcine insulin, etc.); 4) Those who have had severe allergic reactions (such as anaphylactic shock, angioedema) or have a clear history of allergy to two or more different chemical structures of drugs；
3. Known to have alpha-1 antitrypsin deficiency;
4. Severe cognitive impairment: Patients with a score of ≥ 2 on the NIHSS scale for the 1a level of consciousness;
5. Brain CT or MRI indicating large-scale anterior circulation cerebral infarction (the infarction area exceeding one-third of the territory supplied by the middle cerebral artery);
6. Stroke with rapid improvement of symptoms after informed consent, or suspected acute ischemic symptoms caused by other reasons;
7. Those preparing for or having undergone endovascular treatment;
8. Since the onset of this illness, the following drugs with neuroprotective effects have been administered: commercially available edaravone, edaravone-berclor, butylphthalide, human urokinase (Ureklin), pancreatic kallikrein, citicoline, nimodipine, ganglioside, apomorphine, brain glycoprotein, fasudil, compound brain peptide ganglioside, piracetam, oralacetam, cattle serum albumin injection, cattle serum protein extract injection, ginkgo biloba lactone injection, ginkgo diterpene gluconate injection, glutaric acid injection, blood clotting soft capsules, and injections containing any one or more of the following Chinese herbal ingredients: Ligusticum chuanxiong, Salvia miltiorrhiza, Rhodiola rosea extracts；
9. Severe hypertension: After using antihypertensive drugs before random administration, the systolic blood pressure remained ≥ 185 mmHg or the diastolic blood pressure remained ≥ 110 mmHg;
10. Within the 7 days prior to screening, any angiotensin-converting enzyme inhibitor (ACEI: captopril, lisinopril, etc.) was used;
11. During the trial, the plan is to use angiotensin-converting enzyme inhibitors (ACEI: captopril, lisinopril, etc.)；
12. Cases where systolic blood pressure (SBP) was less than 100 mmHg or mean arterial pressure (MAP) was less than 65 mmHg occurred before random grouping after the onset of stroke symptoms; Note: MAP = DBP + [1/3 (SBP - DBP)] (measured using an non-invasive blood pressure cuff device);
13. Patients with active severe infections who require systemic anti-infective treatment;
14. Severe renal dysfunction: Serum creatinine > 2 times the upper limit of normal value or creatinine clearance rate < 30 mL/min (Cockcroft-Gault formula), or known renal failure, uremia and other severe renal dysfunction diseases; (Note: Cockcroft-Gault formula: ① For males: CLcr (mL/min) = [140 - Age (years)] × Weight (kg) / [0.814 × Serum creatinine (μmol/L)]; ② For females: CLcr (mL/min) = { [140 - Age (years)] × Weight (kg) / [0.814 × Serum creatinine (μmol/L)] } × 0.85)；
15. Severe liver dysfunction: ALT or AST is more than 3 times the upper limit of the normal range, or other known liver diseases such as liver failure, cirrhosis, portal hypertension (esophageal varices), active hepatitis, etc.;
16. Patients with a heart function rating of grade II or above (according to the New York Heart Association (NYHA) heart function classification) or those with a history of congestive heart failure;
17. Patients with concurrent malignant tumors or those undergoing anti-tumor treatment;
18. Pregnant women, lactating women, or those planning to become pregnant;
19. Those who have a history of epilepsy or experienced epileptic-like symptoms during a stroke, or those with severe mental disorders, mental impairments, intellectual disabilities or dementia;
20. Those suspected or confirmed to have alcohol dependence, or who consumed more than 3 units of alcohol (for men) or 2 units (for women) within 24 hours before the onset of the disease (1 unit = 360 mL of beer or 45 mL of 40% alcohol liquor or 150 mL of wine);
21. Those who have participated in other drug or non-drug clinical studies within 3 months prior to signing the informed consent form, or are currently involved in other clinical studies;
22. Those with severe systemic diseases and an expected survival period of less than 90 days;
23. Those who cannot tolerate venipuncture or experience dizziness or fainting when standing up, or those who are unwilling to receive multiple intramuscular injections for administration;
24. Patients considered by the researchers to be unsuitable for participating in this clinical study.

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 320 (Estimated)
Dates: Start 2026-01-19 (Actual); Primary Completion 2026-10-31 (Estimated); Study Completion 2026-12-31 (Estimated)

PRIMARY OUTCOMES:
modified rankin scale (mRS) score ≤ 1 | Day 90 after randomization

SECONDARY OUTCOMES:
The modified Rankin Scale (mRS) scores at 90 days after stroke | 90 days after stroke onset
The proportion of participants with a modified Rankin Scale (mRS) score of 0-2 at 30、90 days after stroke onset | 30、90 days after stroke onset
The proportion of participants with a modified Rankin Scale (mRS) score of 0-1 at 30 days after stroke onset | 30 days after stroke onset
The change of the National Institutes of Health Stroke Scale (NIHSS) score from baseline at 14 days after stroke onset | Baseline, 14 days after stroke onset
The proportion of Barthel Index (BI) scores ≥95 at 30 days and 90 days after stroke onset | 30 days and 90 days after stroke onset

OTHER OUTCOMES:
Incidence of adverse events (AE) | From the time of administration to day 90
Incidence of serious adverse events (SAE) | From the time of administration to day 90
All-cause mortality | From the time of administration to day 90

CONTACTS AND LOCATIONS:
Overall Officials: Yun Xu, professor, Principal Investigator — The Affiliated Nanjing Drum Tower Hospital of Nanjing University Medical School
Locations (1):
- Nanjing Drum Tower Hospital, Nanjing, Jiangsu, China

IPD SHARING:
Plan to Share IPD: No